CLINICAL TRIAL: NCT03221101
Title: Home Non Invasive Ventilation Versus Long Term Oxygen Therapy Alone in COPD Survivors After Acute Hypercapnic Respiratory Failure. A French Multicenter Randomized Controlled Trial
Brief Title: Home Non Invasive Ventilation for COPD Patients
Acronym: NIVOLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Collaborators: ADIR Association (Other)
Responsible Party: Principal Investigator, BOUCHRA LAMIA, Professor of medecine, pulmonology. MD, MPH, PhD, University Hospital, Rouen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-AO1276-39 2010/080/HP; CPP-SC 010/2013 (Other: Rouen University, Normandy France)
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Term Oxygen Therapy alone (No Intervention): Long Term oxygen therapy is prescribed according to the guidelines
- Non invasive ventilation (Active Comparator): Home non invasive ventilation is prescribed with the following settings
  * PS mode
  * IPAP according to clinical and hemodynamic tolerance
  * EPAP according to air trapping
  * RR around 12/ min.
  * LOT for SaO2 > 90%
  * Monitoring with capnometry for settings validation
  Interventions: Device: Home ventilator

INTERVENTIONS:
Device: Home ventilator
  Arms: Non invasive ventilation

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) patients are more likely to develop acute hypercapnic respiratory failure. In the acute phase, non invasive ventilation has been shown to improve mortality and reduce intubation rate. Few studies are available about long term benefits of home non invasive ventilation in COPD patients with chronic hypercapnic respiratory failure who survived after an acute episode. The purpose of this study is to determine whether home non invasive ventilation can reduce recurrent acute hypercapnic respiratory failure in COPD patients who survived an acute hypercapnic respiratory failure episode treated by non invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who survived after an acute episode of hypercapnic respiratory failure
* patients weaned from ventilation ( non invasive ventilation or mechanical ventilation) prescribed for acute episode since at least five days with following arterial blood gas : pH > 7.35 and PCO2 > = 45 mmHg

Exclusion Criteria:

* severe obstructive sleep apnea ( DI > 30/h)
* Non COPD cause of respiratory failure
* Serious comorbidity
* Adverse psychological status

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2011-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
acute hypercapnic respiratory failure episode | up to 24 months
  first episode of acute hypercapnic respiratory failure episode requiring hospitalization

SECONDARY OUTCOMES:
acute hypercapnic respiratory failure episode rate | up to 24 months
pulmonary function test | at one month and every six months up to 24 months
Six Minute Walk Distance | at one month and every six months up to 24 months
Quality of life | at one month and every six months up to 24 months
Heart function | at one month and every six months up to 24 months
  left and right heart function assessed using echocardiography
Cost effectiveness | at one month and every six months up to 24 months
mortality | at one month and every six months up to 24 months
arterial blood gas | at one month and every six months up to 24 months

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH Dieppe, Dieppe
  - CH Elbeuf, Elbeuf
  - Le Havre, Jacques Monod Hospital, Montivilliers
  - CHU de Rouen, Rouen